CLINICAL TRIAL: NCT00978770
Title: Neo Comice Pilot; Efficacy of Advanced Semi-automated Functional Magnetic Resonance (MR) Imaging in the Early Prediction of Response of Locally Advanced Breast Cancer to Neoadjuvant Chemotherapy
Brief Title: MRI in Predicting Early Response to Chemotherapy in Patients With Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Clinical Trials Unit, Scotland (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: CCTU-Neo-COMICE; CDR0000649054 (Registry Identifier: PDQ (Physician Data Query)); ISRCTN42613663; EU-20968
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2009-09

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy; Magnetic Resonance Spectroscopy

INTERVENTIONS:
Drug: systemic chemotherapy
Procedure: diffusion-weighted magnetic resonance imaging
Procedure: dynamic contrast-enhanced magnetic resonance imaging
Procedure: magnetic resonance spectroscopic imaging
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Diagnostic procedures such as MRI scans may help predict early response to treatment in patients with breast cancer undergoing chemotherapy.

PURPOSE: This phase II trial is studying MRI in predicting early response to chemotherapy in patients with locally advanced breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the technical feasibility of using MRI in a multicenter setting using the most commonly available magnetic resonance (MR) systems (i.e., is the trial able to scan patients to a specific protocol, using different types of MRI machine) measured by the number of MRI scans not completed to technical specifications (i.e., incorrect sequences or incomplete scans) or trial protocol (i.e., scans not completed or completed at the wrong time).
* To determine how reliably the imaging data can be analyzed in a centralized, semi-automated manner (i.e., can MRI data be reliably transferred from different centers and analyzed using software based in the center for MR investigations at the University of Hull) measured by the number of cases where automated data analysis of completed MRI scans was not possible (i.e., data could not be analyzed at all or data required manual analysis).

OUTLINE: This is a multicenter study.

Patients undergo magnetic resonance imaging (MRI) scans at baseline, 4-7 days after beginning after the first course of chemotherapy, at the end of their second course of chemotherapy, and at the end of their fourth course of chemotherapy (first regimen). MRI techniques may include dynamic contrast-enhanced, diffusion-weighted, and spectroscopic.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed, histologically proven breast cancer

  * Stage T2-4B, N0-3C, and M0 disease
  * Locally advanced primary disease
* Underwent both x-ray mammography and breast ultrasound scanning during the current treatment episode
* Scheduled for neoadjuvant chemotherapy

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Medically stable
* No renal failure
* No serious breast trauma within the past 3 months
* No known allergic reaction associated with previous administration of a paramagnetic contrast agent
* No known contraindication to magnetic resonance (MR) scanning

  * Must pass the normal safety requirements of MR, particularly pacemakers and cardiac defibrillators
  * No disability preventing MR scanning in the prone position
  * No body habitus incompatible with MR system entry

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy
* No prior surgery or radiotherapy for cancer in the ipsilateral breast

  * More than 4 months since prior surgery to the ipsilateral breast for benign breast disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-08; Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Failed scan rate (i.e., the number of scans that failed protocol) grouped by cause, including patient refusal, protocol violation in timing, major errors in scan protocols, and minor errors in scan protocol
Failed automated MRI-scan data-analysis rate (i.e., number of scans that required manual reading and number of protocol-compliant scans that were unreadable, subdivided according to whether the scans were technically compliant or not)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay W. Turnbull, MD, Principal Investigator — Hull Royal Infirmary
Locations (1):
- Cactus Clinical Trials Unit, Hull, England, United Kingdom